CLINICAL TRIAL: NCT06610916
Title: Faisability and Efficacity of the Reinforced Communautary Support Program (PARC) on the Complications of Chemsex
Acronym: E-PARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP231561; IDRCB: 2024-A00651-46 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Chemsex; Addiction; Infections; Sexual Disorder, Physiological
Keywords: chemsex; MSM; addiction; sexual health; HIV
MeSH Terms: conditions — Chemsex; Behavior, Addictive; Infections; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reinforced Communautary Support Program (PARC) (Experimental): Participants will complete the initial self-questionnaire collecting baseline socio-demographic, clinical characteristics, and all intermediate effectiveness outcome criteria "before". Concurrently with their participation in the program, they will complete various intermediate effectiveness evaluation questionnaires ("after") at 3 months (end of PARC) and 6 months (Post-PARC). Healthcare professionals running the PARC program will also complete questionnaires related to implementation indicators throughout the patients' course (Adoption, Implementation, Maintenance).
  Qualitative interviews will be conducted with patients and relevant healthcare professionals to explore barriers and drivers to the optimal deployment of the PARC program and to examine each of the Reach, Adoption, Implementation, Maintenance indicators through an organizational approach
  Interventions: Other: Reinforced Communautary Support Program (PARC)

INTERVENTIONS:
Other: Reinforced Communautary Support Program (PARC) — Participants will complete the initial self-questionnaire collecting baseline socio-demographic, clinical characteristics, and all intermediate effectiveness outcome criteria "before". Concurrently with their participation in the program, they will complete various intermediate effectiveness evaluation questionnaires ("after") at 3 months (end of PARC) and 6 months (Post-PARC). Healthcare professionals running the PARC program will also complete questionnaires related to implementation indicators throughout the patients' course (Adoption, Implementation, Maintenance).
  Qualitative interviews will be conducted with patients and relevant healthcare professionals to explore barriers and drivers to the optimal deployment of the PARC program and to examine each of the Reach, Adoption, Implementation, Maintenance indicators through an organizational approach

SUMMARY:
The complications associated with chemsex concern infectious disease specialists, addiction specialists, and public authorities. Chemsex is defined among men who have sex with men (MSM) and trans and non-binary individuals participating in gay hookup networks due to their specific psychological, sexual, and social characteristics. The drugs used in France are cathinones (3MMC), GBL, and methamphetamine, administered orally, nasally, rectally, and intravenously (""slam"").

Building on change models and health education theories, the teams at 190 and Spot Beaumarchais (AIDES) have created, within their shared facilities, the Parcours d'Accompagnement Renforcé Communautaire (PARC), a multidisciplinary and community-based program providing comprehensive care for chemsex complications. The program aims to achieve clinical benefits:

* Reducing addiction symptoms
* Decreasing somatic, psychiatric, and social risks related to chemsex
* Exploring and addressing the determinants of consumption and complications, especially psychological and psychiatric
* Improving social connections
* Maintaining life and professional goals
* Perceiving or creating new types of connections between men
* Resuming physical activity
* Improving self-esteem
* Finding a satisfying and fulfilling sexuality
* Enhancing overall quality of life

The goal of this study is to ensure that the PARC program, as designed, reaches its target population, is feasible, sustainable, at an acceptable cost, and improves the conditions of the population accessing it throughout the course. Thus, in the medium term, this study will identify all success factors for deploying such a program and build a toolkit for its dissemination to other regions with similar issues but somewhat different contexts.

The primary objective is to evaluate the feasibility of the PARC program in terms of implementation by measuring patient adherence to the program.

The primary outcome measure is the rate of patients who completed the follow-up in the PARC program compared to the number of patients who started the PARC program (at least the inclusion visit) over 18 months. A patient is considered adherent if they have attended at least one of each type of workshop offered during the first month AND continued to attend at least 4 workshops and 2 consultations per month during months 2 and 3.

The secondary objectives are:

1. To evaluate the feasibility of the PARC program in terms of implementation, using the RE-AIM methodology (Glasgow):

   * Reach: Does the included patient population accurately represent the target population? Does patient loss represent the most vulnerable patients?
   * Intermediate Effectiveness at 3 months: (self-administered questionnaires)
   * Overall quality of life
   * Addiction criteria
   * Somatic complications
   * Social life
   * Sexual quality of life
   * Adoption of the intervention by professionals: Do addiction networks, CeGIDD, CSAPA, and city doctors refer their patients to the PARC program?
   * Implementation of the intervention: Has the program evolved from the beginning to the end of the study? Have there been adaptations?
   * Maintenance or sustainability: Is the financial model of the program sustainable and does it ensure a return on investment by analyzing the cost of care?
2. To identify contextual factors that are facilitators or barriers to optimal implementation and effectiveness. (qualitative analysis)

The expected sample size is 60 patients included over a period of 18 months. Each patient will be included for a duration of 6 months, and the study will last for 24 months.

Once included, participants will complete the initial self-questionnaire collecting baseline socio-demographic, clinical characteristics, and all intermediate effectiveness outcome criteria ""before"". Concurrently with their participation in the program, they will complete various intermediate effectiveness evaluation questionnaires (""after"") at 3 months (end of PARC) and 6 months (Post-PARC). Healthcare professionals running the PARC program will also complete questionnaires related to implementation indicators throughout the patients' course (Adoption, Implementation, Maintenance).

Qualitative interviews will be conducted with patients and relevant healthcare professionals to explore barriers and drivers to the optimal deployment of the PARC program and to examine each of the Reach, Adoption, Implementation, Maintenance indicators through an organizational approach

DETAILED DESCRIPTION:
At 190, a community sexual health center in Paris, more than one in five patients engage in chemsex. The complications associated with chemsex concern infectious disease specialists, addiction specialists, and public authorities. These complications are somatic, addiction-related, sexual, and psychiatric. They are both severe and frequent (estimated difficulties between 30% and 50% of users) and there is no effective treatment for stimulant addiction. The drugs used in France are cathinones (3MMC), GBL, and methamphetamine, administered orally, nasally, rectally, and intravenously ("slam"). According to the European Chemsex Forum, drug use in a sexual context is not necessarily chemsex. Chemsex is defined among men who have sex with men (MSM) and trans and non-binary individuals participating in gay hookup networks due to their specific psychological, sexual, and social characteristics.

A community-based program (Getting Off - Los Angeles) combining group therapy and contingency management is currently the only known intervention that has shown potential benefits in reducing consumption and HIV-related risks among methamphetamine-using chemsex practitioners (Reback et al. 2014; Blair et al. 2022). This program requires multiple practitioners and cross-disciplinary knowledge in community and medical care, psychology, and sexology. Structures like CSAPA (addiction care centers) or CeGIDD (sexual health centers) lack this multidisciplinary approach, and access to comprehensive care is limited due to the caregivers' lack of knowledge and the users' apprehension about judgment regarding sexuality and drugs.

Building on change models and health education theories, the teams at 190 and Spot Beaumarchais (AIDES) have created, within their shared facilities, the Parcours d'Accompagnement Renforcé Communautaire (PARC), a multidisciplinary and community-based program providing comprehensive care for chemsex complications. The program aims to achieve clinical benefits in several areas:

* Reducing addiction symptoms
* Decreasing somatic, psychiatric, and social risks related to chemsex
* Exploring and addressing the determinants of consumption and complications, especially psychological and psychiatric
* Improving social connections
* Maintaining life and professional goals
* Perceiving or creating new types of connections between men
* Resuming physical activity
* Improving self-esteem
* Finding a satisfying and fulfilling sexuality
* Enhancing overall quality of life

Since the PARC program was recently implemented at 190, the goal of this study is to assess its effectiveness through the lens of its implementation. Using the RE-AIM implementation evaluation model, the E-PARC study will assess the program's transferability to the French context and its effectiveness on intermediate indicators, without comparison to a control group. The aim is to ensure that the PARC program, as designed, reaches its target population, is feasible, sustainable, at an acceptable cost, and improves the conditions of the population accessing it throughout the course. The goal is not to demonstrate that all centers should adopt this program, but to show that this specific expert program best fulfills its function for a vulnerable population-due to its risk behaviors and the lack of current care-by addressing each of its specific needs. This is to ensure that the PARC program is known, recognized, and strengthened to receive as many patients as possible outside of care or referred by healthcare professionals encountering chemsex practitioners. PARC is currently the only program that effectively supports chemsex practitioners, is multi-component, based on evidence-based medicine, led by the leading French gay community sexual health center, and recognized by the gay community. This program encompasses all leverage factors necessary for optimal care for the target population.

Thus, in the medium term, this study will identify all success factors for deploying such a program and build a toolkit for its dissemination to other regions with similar issues but somewhat different contexts.

The primary objective is to evaluate the feasibility of the PARC program in terms of implementation by measuring patient adherence to the program.

The primary outcome measure is the rate of patients who completed the follow-up in the PARC program as described in the model compared to the number of patients who started the PARC program (at least the inclusion visit) over 18 months.

The secondary objectives are:

1. To evaluate the feasibility of the PARC program in terms of implementation, using the RE-AIM methodology (Glasgow):

   * Reach: Does the included patient population accurately represent the target population? Does patient loss represent the most vulnerable patients?
   * Intermediate Effectiveness at 3 months:
   * Overall quality of life
   * Addiction criteria
   * Somatic complications
   * Social life
   * Sexual quality of life
   * Adoption of the intervention by professionals: Do addiction networks, CeGIDD, CSAPA, and city doctors refer their patients to the PARC program?
   * Implementation of the intervention: Has the program evolved from the beginning to the end of the study? Have there been adaptations?
   * Maintenance or sustainability: Is the financial model of the program sustainable and does it ensure a return on investment by analyzing the cost of care?
2. To identify contextual factors that are facilitators or barriers to optimal implementation and effectiveness.

The secondary outcome measures are:

1. The implementation:

   * Reach:
   * Number of patients offered the program
   * Number and reasons for refusals
   * Intermediate Effectiveness at 3 months:
   * Overall quality of life: WHOQOL26
   * E-PARC Questionnaire: Impact of chemsex: ad hoc chemsex complications questionnaire
   * All substances addiction: Brief Addiction Monitor (Cacciola)
   * Craving: Craving Questionnaire (Weiss)
   * Social life: Multidimensional Scale of Perceived Social Support (Zimet)
   * Sexual quality of life: The New Sexual Satisfaction Scale (Štulhofer)
   * Adoption:
   * Number of primary care professionals referring patients to the PARC program, original structure of these professionals
   * Number of non-healthcare professionals referring individuals to the PARC program, original structure
   * Mapping of the patient referral network, comparison to the community and addiction network
   * Implementation:
   * Number of workshops attended by each patient
   * Frequency of visits to the PARC
   * Number of planned/actual visits
   * Most and least attended workshops
   * Evolution of the program structure during the study
   * Maintenance:
   * Cost for funders for one year of PARC implementation
   * Cost per patient followed
2. The barriers and Facilitators:

   * Contextual elements identified through qualitative analysis (Michie) with professionals and users

The eligibility criteria are:

* Adult men engaging in chemsex seeking care:
* Men who have sex with other men and/or non-binary individuals, trans men or women associated with gay sexual networks
* Engaging in chemsex (as defined by the European Chemsex Forum and having consumed at least twice a cathinone and/or methamphetamine and/or GHB/GBL)
* Seeking care for chemsex
* Referred to the PARC program with the goal of reducing or stopping consumption
* Not opposed to data collection for this study
* Uncontrolled somatic or psychiatric conditions
* Refusal to participate

Eligible patients will be invited to participate in the E-PARC study (information sheet provided by investigators, collection of non-opposition). The expected sample size is 60 patients included over a period of 18 months. Each patient will be included for a duration of 6 months, and the study will last for 24 months.

Once included, participants will complete the initial self-questionnaire collecting baseline socio-demographic, clinical characteristics, and all intermediate effectiveness outcome criteria "before." Participants will then enter the PARC program. Concurrently with their participation in the program, they will complete various intermediate effectiveness evaluation questionnaires ("after") at 3 months (end of PARC) and 6 months (Post-PARC). Healthcare professionals running the PARC program will also complete questionnaires related to implementation indicators throughout the patients' course (Adoption, Implementation, Maintenance).

Qualitative interviews will be conducted with patients and relevant healthcare professionals to explore barriers and drivers to the optimal deployment of the PARC program and to examine each of the Reach, Adoption, Implementation, Maintenance indicators through an organizational approach. These interviews will occur throughout the study and will be conducted by a researcher trained in human and social sciences.

The adherence rate to the program will be calculated as follows:

A patient is considered adherent if they have attended at least one of each type of workshop offered during the first month AND continued to attend at least 4 workshops and 2 consultations per month during months 2 and 3.

The adherence rate is calculated as: number of patients considered adherent / Number of patients included Descriptive analyses of collected variables for assessing implementation and all these domains will be conducted: using frequencies (percentages) or medians (interquartile ranges), as appropriate, and reporting the number of missing data. A mapping analysis of patient flows will be performed. Results of intermediate effectiveness outcome measures before and after will be compared using the Wilcoxon signed-rank test for paired samples-non-parametric-with a significance threshold of p < 0.05. All analyses will be conducted using SAS® and by the URC of Robert Debré Hospital to ensure quality assurance.

ELIGIBILITY:
Inclusion Criteria:

* MSM and/or non-binary individuals, trans men or women associated with gay sexual networks
* Engaging in chemsex (as defined by the European Chemsex Forum and having consumed at least twice a cathinone and/or methamphetamine and/or GHB/GBL)
* Seeking care for chemsex
* Referred to the PARC program with the goal of reducing or stopping consumption
* Not opposed to data collection for this study
* Uncontrolled somatic or psychiatric conditions

Exclusion Criteria:

* Refusal to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who completed the follow-up in the PARC program as described in the model compared to the number of patients who started the PARC program (at least the inclusion visit) | 18 months
  Rate of patients who completed the follow-up in the PARC program as described in the model compared to the number of patients who started the PARC program (at least the inclusion visit)

CONTACTS AND LOCATIONS:
Overall Officials: Michel OHAYON, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Le 190 - Centre de Santé Sexuelle / CeGIDD, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided